CLINICAL TRIAL: NCT03136471
Title: Natural Experiments of the Impact of Population-Targeted Health Policies to Prevent Diabetes and Its Complications
Brief Title: Impact of CMS Reimbursement Policy Supporting Care Coordination in Louisiana
Status: Completed | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 16-906810
Record Dates: First submitted 2017-03-24; First posted 2017-05-02 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2; Chronic Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- EMR data extraction: EMR Data extraction from the Louisiana Clinical Data Research Network (LaCDRN). The Louisiana Clinical Data Research Network (LaCDRN) data will be requested, including patients' records of pharmacy, inpatient, outpatient and lab results from January 01, 2016 to December 31, 2021. It is a retrospective data analysis without interaction with any participants. All data is de-identified and the study participants will not be contacted in any way.
  Inclusion criteria: Patients with type 2 diabetes, whose age>=18 years old will be extracted from database of LaCDRN.
  Exclusion criteria: Patients without type 2 diabetes or age<18 years old.
- Healthcare Professionals: Healthcare professionals (physician, nurse) will be randomly selected from LaCDRN partner health system. An email will be distributed to the registered clinicians at partner health systems.
  Inclusion criteria: physicians and nurses who treat diabetes patients and work at clinic settings within LaCDRN network and consent to participate the study.
  Exclusion criteria: physicians and nurses who do not treat diabetes patients or not work at clinic settings within LaCDRN network; refuse to participate the study.
- Patients for Qualitative Study: Patients with diabetes who are a members of Diabetes Advisory Group or partner LaCDRN health system will be contacted via email, letter or phone call.
  Inclusion criteria:
  * Diabetes patients who consent to participate the study.
  * Age 65+;
  * Diagnosis code for diabetes in the last 2 years;
  * Diagnosis code for at least one additional chronic condition in the last 2 years.
  Exclusion criteria: age<65; patient with diabetes without other chronic conditions.
- LaCDRN partner health system's medical directors: Face-to-face semi-structured interviews will be used to explore organizational cultures, their social architecture, resources, capacity, communication networks, assess barriers, and refine the data collection for the assessing the RE-AIM framework. The one time interview will take 1 hour. A 10 minutes questionnaire of Diabetes care coordination readiness assessment (DCCRA) will be emailed to them annually during entire 5 years of study period.
- PROMIS® survey: Patients for PROMIS® survey (National Institutes of Health's Patient-Reported Outcome Measurement Information System Global Health Measures). Patients will be administered the surveys at the point-of-care visit (in exam rooms) using REACHnet's tablet-based application.
  Inclusion criteria:
  * All patients age 18+ who registered at REACHnet.
  * Able to provide informed consent
  Exclusion criteria: patients who do not provide inform consent or age<18 years old.
- PACIC+ survey: Patients for PACIC+ survey (Group Health Research Institute's Patient Assessment of Care for Chronic Conditions+). Patients will be administered the surveys at the point-of-care visit (in exam rooms) using REACHnet's tablet-based application.
  Inclusion criteria:
  * All patients age 18+ with a Diabetes diagnosis and who registered at REACHnet.
  * Able to provide informed consent
  Exclusion criteria: patients who do not provide inform consent or without diabetes diagnosis or age<18 years old
- Telehealth Services using HCPCS/CPT for COVID-19 Patients: Study population with versus without telehealth services. Telehealth services using the HCPCS/CPT codes will be defined in the following categories: Medicare telehealth visits (CPT codes: 99201-99215; HCPCS codes: G0425-G0427, G0406-G0408), virtual check-in (HCPCS codes: G2010, G2012), and e-visits (CPT codes: 99421-99423, HCPCS codes: G2061-G2063). Propensity score-matching will be used to ensure comparison groups are comparable at baseline.

SUMMARY:
Investigators propose to use a natural experiment design to examine the impacts of the new CPT code (99490) for chronic care management on health outcomes. The Investigators will collaborate with partners in the Louisiana Clinical Data Research Network (LaCDRN) who serve more than 90,000 patients with type 2 diabetes mellitus in Louisiana to examine impacts of the CMS reimbursed care coordination. Now, LaCDRN is renamed as Research Action for Health Network (REACHnet). Patient and stakeholder engagement will be planned and implemented across all phases of this natural experiment. This project will examine outcome differences created by the policy change in a natural experiment framework. The analyses will utilize the RE-AIM framework to identify the critical elements of the programs that will enhance the reach, effectiveness, adoption, implementation, and maintenance of these strategies in the diverse LaCDRN diabetes populations.

PCORI Proposal COVID-19- Related Enhancement for Existing Research:

The proposed enhancement will contribute timely information to address two important implications of the coronavirus pandemic:

1. Disparities in continuity of care and
2. Health systems' responsiveness in terms of telehealth delivery for high risk populations.

The enhancement builds upon our current project by further examining effects of CMS payment innovations to expand remotely delivered care. Our proposed study is a rapid assessment of telehealth services, using an existing "learning health system" infrastructure to provide timely, actionable evidence to inform telehealth service provision during the pandemic and recovery.

DETAILED DESCRIPTION:
The first aim is to evaluate the barriers and facilitators for the RE-AIM dimensions as related to the new CMS chronic care management code overall and within each of the health systems. The qualitative study will be used. Focus group interview will be conducted among patients, healthcare professionals and stakeholders. A variety of qualitative techniques will be used to collect data using key informant interviews among organization leaders of LaCDRN partners to assess the organizational cultures, their social architecture, resources, capacity, and communication networks. Face-to-face semi-structured interviews will be used to explore these domains, assess barriers, and refine the data collection for the assessing the RE-AIM framework. Further, semi-structured interviews will provide data to inform the refinement of study outcomes and ensure organizational, cultural, and health-literacy appropriateness. Focus groups will be audiotaped with the written consent of each participant, and each tape will be transcribed verbatim and transcripts will be reviewed and edited by the facilitators for accuracy. Inter-coder reliability will be examined. Interview transcripts will be imported into NVivo 10 software (QSR International, Burlington, MA). Codes and concepts identified in preliminary review will be refined, extended, and cross-referenced. Coded texts will be structured into taxonomies and transformed into a matrix format so that responses and concepts can be compared across respondent groups. Finally, taxonomies and matrices will be summarized by similarities and contrasts to form overarching themes and dimensions. We will use an iterative technique until theoretical saturation, the point at which no additional major themes emerge, is reached. Diabetes care coordination readiness assessment will be conducted with LaCDRN partner health system's medical directors (organizational).

The second one is the health and economic impacts of the NFFCCM to improve health outcomes: glycemic control, CVD risk reduction, medication adherence, patient-reported outcomes (PRO), and health care utilization. Data extraction from the REACHnet. De-identified data from EMR includes birth year, gender, race, state of residency, zip-codes, medical history, lab results and prescriptions. All data comply with the Health Insurance Portability and Accountability Act (HIPAA).

This proposed research is significant because it is the first natural experiment to test an ongoing CMS reimbursement policy on diabetes care in Louisiana. The study questions and study outcomes will be patient-centered, and will generate urgently needed data on effective, practical, and sustainable population-targeted strategies aimed at reducing diabetes-related disease burden in Medicare-eligible populations. Further dissemination and scale-up efforts will create large return on multiple health systems and non-CMS populations.

PCORI Proposal COVID-19- Related Enhancement for Existing Research Aims:

Aim1: Examine facilitators and barriers to uptake, adoption, and implementation of telehealth services among Medicare patients with diabetes from health systems', providers' and patients' perspectives. With the substantial increase in telehealth encounters starting in early March 2020, we hypothesize disparities in adoption and implementation of telehealth at health system, provider and patient levels. For example, our current project has identified significant variations in NFFCCM implementation across three health systems in Louisiana. For the enhancement, we intend to examine variations in health systems' implementation of Medicare-reimbursable telehealth services, which may not mirror the variations we observed for NFFCCM given the dramatically different context of the current pandemic.

Aim 2: Compare diabetes control and continuity of care between patients with and without utilization of telehealth. We hypothesize better diabetes management among Medicare patients with telehealth versus without.

ELIGIBILITY:
Healthcare professionals (physician, nurse) will be randomly selected from LaCDRN partner health system.

* Inclusion criteria: physicians and nurses who treat diabetes patients and work at clinic settings within LaCDRN network and consent to participate the study.
* Exclusion criteria: physicians and nurses who do not treat diabetes patients or not work at clinic settings within LaCDRN network; refuse to participate the study.

Patients for qualitative study:

* Inclusion criteria: Diabetes patients who consent to participate the study; Age 65+; Diagnosis code for diabetes in the last 2 years; Diagnosis code for at least one additional chronic condition in the last 2 years.
* Exclusion criteria: age<65; patient with diabetes without other chronic conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes Healthcare professionals who treat diabetes patients, medical directors at Louisiana Clinical Data Research Network (LaCDRN) affiliated clinics, patients with diabetes, patients who are registered with REACHnet, and medical records from LaCDRN affiliated clinics.
Sampling Method: Probability Sample
Enrollment: 22242 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in use of CMS care coordination reimbursement code over 5 years | 5 years
  Over 5 years the utilization of the CMS care coordination reimbursement code will be analyzed to see if there is any change in how often the code is used.
Change in glycemic control over 5 years | 5 years
  Over 5 years diabetes patients extracted from the EMR will be analyzed to see if patients are able to achieve glycemic control by having a Hemoglobin A1c <7% and maintain staying below 7.0%.
Change in healthcare utilization over 5 years | 5 years
  Records from the EMR will be assessed by counting the number of outpatient visits, number of inpatient visits, and number of emergency room visits, to determine if there has been a change in the utilization of the healthcare system.
Change in patient satisfaction over 5 years | 5 years
  Patients registered in REACHnet, diagnosed with Type 2 diabetes, and complete the PACIC+ survey will be analyzed to see if there is a change in patient satisfaction over 5 years.
Change in status of received diabetes care over 5 years | 5 years
  Patients registered in REACHnet, diagnosed with Type 2 diabetes, and complete the PACIC+ survey will be analyzed to see if there is a change in the patient's status of received diabetes care over 5 years.
Change in patient reported physical health over 5 years | 5 years
  Patients registered in REACHnet and complete the PROMIS survey will be analyzed to see if there is a change in patient reported physical health score over 5 years.
Glycemic Control (HbA1c) for Telehealth visits for COVID-19 patients | Baseline, post-baseline period within 12 months
  Measured before and within 12 months after 03/06/2020

CONTACTS AND LOCATIONS:
Overall Officials: Lizheng Shi, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Walker B, Stoecker C, Shao Y, Nauman E, Kabagambe EK, Shi L. Predictors of Telehealth Utilization and Subsequent Inpatient Stays and Emergency Visits During the COVID-19 Pandemic Among Patients with Type 2 Diabetes: Evidence from Louisiana. Telemed J E Health. 2024 Jan;30(1):278-283. doi: 10.1089/tmj.2022.0509. Epub 2023 Jul 3. PMID 37405746